CLINICAL TRIAL: NCT03471455
Title: A Pilot Study to Assess The Therapeutic Effectiveness Of Isotretinoin In Preventing Recurrences In Chronic Recurrent Dermatophytosis
Brief Title: Isotretinoin In Preventing Recurrences In Chronic Recurrent Dermatophytosis
Acronym: ISORD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Tarun Narang, ASSISTANT PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT/IEC/2017/850
Record Dates: First submitted 2018-02-06; First posted 2018-03-20 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Tinea
MeSH Terms: conditions — Tinea | interventions — Isotretinoin; Terbinafine; Itraconazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Terbinafine alone (Active Comparator): Patients of recurrent dermatophytosis (recurrent episodes for more than 6 months) will receive oral terbinafine 250 mg once a day for 4 weeks.
  Interventions: Drug: Terbinafine
- Terbinafine plus isotretinoin (Active Comparator): Patients of recurrent dermatophytosis (recurrent episodes for more than 6 months) will receive oral terbinafine 250 mg once a day for 4 weeks and oral isotretinoin 20 mg/ day for 6 months.
  Interventions: Drug: Isotretinoin; Drug: Terbinafine
- Itraconazole only (Active Comparator): Patients of recurrent dermatophytosis (recurrent episodes for more than 6 months) will receive oral itraconazole 200 mg twice a day for 4 weeks.
  Interventions: Drug: Itraconazole 200 mg
- Itraconazole plus isotretinoin (Active Comparator): Patients of recurrent dermatophytosis (recurrent episodes for more than 6 months) will receive oral itraconazole 200 mg twice a day for 4 weeks and oral isotretinoin 20 mg/ day for 6 months.
  Interventions: Drug: Isotretinoin; Drug: Itraconazole 200 mg

INTERVENTIONS:
Drug: Isotretinoin — Patients of recurrent dermatophytosis will receive terbinafine or itraconazole , either alone or in combination with oral isotretinoin
  Arms: Itraconazole plus isotretinoin; Terbinafine plus isotretinoin
Drug: Terbinafine — Patients of recurrent dermatophytosis will receive terbinafine or itraconazole , either alone or in combination with oral isotretinoin
  Arms: Terbinafine alone; Terbinafine plus isotretinoin
Drug: Itraconazole 200 mg — Patients of recurrent dermatophytosis will receive terbinafine or itraconazole , either alone or in combination with oral isotretinoin
  Arms: Itraconazole only; Itraconazole plus isotretinoin

SUMMARY:
This study is a prospective, double blinded, randomized, pilot study to assess the effectiveness of oral low dose isotretinoin in combination with oral terbinafine and itraconazole in preventing recurrences in chronic recurrent dermatophytosis. The recruited patients will be randomized into four treatment arms; oral terbinafine alone and oral itraconazole alone versus oral isotretinoin in combination with each of these two antifungal agents. Randomization will be done using computer generated random number table. The patients in first treatment arm will receive 250 mg of oral terbinafine for 4 weeks, the patients in second treatment arm will receive oral itraconazole 200 mg twice a day for the same duration, while the patients in the third arm will receive oral terbinafine 250 mg once a day for 4 weeks with oral isotretinoin 20 mg once daily and patients in the fourth arm will receive oral itraconazole 200 mg twice a day for 4 weeks with oral isotretinoin 20 mg once daily. In the third and fourth arms, oral terbinafine and oral itraconazole respectively will be stopped after 4 weeks while oral isotretinoin will be continued for 6 months with monthly monitoring of liver function tests and fasting lipid profile.The patients will be followed at monthly intervals for recurrence and treated appropriately.

The primary objective is to evaluate the effectiveness of low dose isotretinoin (20 mg/day) in preventing recurrences in chronic recurrent dermatophytosis by comparing the frequencies of recurrence in patients who are on low dose isotretinoin during the follow up versus those who are not comparing the disease free interval between the four randomized groups at monthly follow up for a total duration of 6 months.

DETAILED DESCRIPTION:
Over the last couple of years, the major concern in dermatophytic infections has been the occurrence of recurrent infections. This, in spite of the patients being treated with gold standard drugs, namely, terbinafine, griseofulvin, and even azoles like itraconazole, in adequate doses. The world is experiencing a menace of recurrent and chronic dermatophyte infections in a magnitude that is unprecedented. Such cases are making up a large proportion of cases seen every day in the outpatient department. To make matters worse, there is as yet, no standard definition of the terms 'çhronic', 'recurrent', or 'resistant' tinea infections, although arbitrary definitions exist, like 'chronic dermatophytosis' being described in lay terms as "patients who have suffered from the disease for more than 6 months to 1 year duration, with or without recurrence, in spite of being treated", and recurrent dermatophytosis being defined as the reoccurrence of the dermatophyte infection within few weeks, after completion of treatment.

Alteration of immune pattern in dermatophytosis The development of antibodies (IgM, IgG, IgA and IgE) to dermatophyte infection seems not to substantially contribute to the elimination of fungal infections because highest antibody levels can be found in patients with chronic fungal infections. Studies by Jones in human volunteers suggested that cell-mediated immunity is the major immunologic defence mechanism in dermatophyte infection.Healthy volunteers infected with T. Mentagrophytes developed cell-mediated immunity resulting in mycologic cure. This was associated with intense inflammation due to T-cell mediated DTH, judging from the trichophytin skin test. A protective immunologic memory was indicated by elimination of T. mentagrophytes on re-inoculation and a continued positive trichophytin test. Impaired cell-mediated immunity in atopic persons is also believed to be the underlying mechanism for an increased susceptibility to T rubrum infections. Patients with allergic bronchial asthma or allergic rhinitis often develop chronic or recurrent fungal infections associated with high immediate-type hypersensitivity (high IgE levels) and low or waning DTH to trichophytin.

Green et al. showed that athymic rats that lack T-cell-mediated immunity could not clear T. mentagrophytes infection in contrast to their genetically matched euthymic control rats.

Chronic dermatophytosis is associated with a depression in cell-mediated immunity to dermatophytes. A selective antigen-specific immunodeficiency may be the underlying factor in such patients, and the continued presence of infecting dermatophytes or residual fungal elements may induce a tolerant state by flooding the host with antigenic material, resulting in a selective loss of cell-mediated immunity. Alternatively, fungal elements may interact with host skin to alter the cytokine milieu such that effective type I immune responses for eliminating organisms are suppressed. In a study done to evaluate immune response in T rubrum onychomycosis and to determine whether immune reactivity or nonreactivity can be a predictor of therapeutic outcome, a double-blind comparison was done of the effects of terbinafine with placebo tablets. Skin tests were performed using trichophytin antigen injected intradermally in the upper left arm. It was found that skin reactivity to trichophytin antigen decreases with increasing disease chronicity. Patients with longstanding disease demonstrated absent or significantly blunted skin reaction to trichophytin antigen compared with patients who had disease for less than 5 years. Patients who were reactive at baseline were the first to become mycologically negative in response to terbinafine treatment, and increases in skin reactivity were related to conversion to negative mycology. Subjects anergic at baseline who converted with treatment had a more favorable outcome overall than persistent nonconverters. It is already known that terbinafine and azoles eliminate the fungal elements and restore cellular immunity resulting in eradication of the oragnisms and cure of the infection. In our study, we plan to analyse if low dose oral isotretinoin has any role to play in the maintenance of the cure achieved by itraconazole by decreasing the number of relapses and whether it leads to an alteration of skin reactivity to trichophytin. If indeed we observe that isotretinoin does, in fact, reduce the number of relapses, it would be interesting to know if there is an immunological basis for this, given that isotretinoin is known to be an immunomodulator.

Probable antifungal Resistance Mechanisms in Dermatophytes In vivo, anti fungal resistance is also correlated with antifungal misuse because patients often fail to finish the full course of treatment. Thus, the inadequate use or dosage of drugs contributes to the failure in eliminating the disease agent completely, encouraging growth of the most resistant strains, which may lead to hard-to-treat fungal infections.

Only few reports have addressed the drug resistance mechanism in dermatophytes, and most of them have been described in T. rubrum. It is noteworthy that resistance to a particular drug can be achieved by more than one mechanism and probably, under certain circumstances, they are activated simultaneously.

Although dermatophytes have powerful metabolic machinery for survival, they have to overcome many pitfalls imposed by the host. Thus, dermatophytes have developed mechanisms that allow them to avoid the host defences such as the immunosuppressive action of fungal mannans that causes reduction of inflammation and phagocytosis. The chemical composition of the cell wall of dermatophytes plays an important role in pathogenicity because of the existing correlation between alteration in the chemical composition of the cell wall, cell dimorphism and virulence.

Probable role of Isotretinoin against dermatophytes Following adherence, successful installation of dermatophytes requires rapid germination of arthroconidia and penetration of hyphae into the stratum corneum. Failure to do so results in elimination by the continuous desquamation of the epithelium. Retinoids act as modulators of epidermal growth and differentiation. Although they normalize proliferation in hyperproliferative epithelia as in psoriasis; in normal epidermis, they promote cell proliferation. Therefore, increased cell turnover in the epidermis may halt the spread of ongoing infection by eliminating the growing dermatophyte. Retinoids are also known to alter terminal differentiation towards a non-keratinizing, metaplastic and mucosa-like epithelium.

Another aspect is the altered glycosylation pattern of normal skin treated with retinoic acid that resembles that of mucosal epithelium with a reduction of tonofilaments, decreased corneocyte cohesiveness, impaired function of the permeability barrier and increased transepidermal water loss. This could thus explain the keratolytic effect of retinoids in hyperkeratotic disorder and could be extrapolated to any probable role of isotretinoin that we see in chronic and recurrent dermatophyte infections.

Once established, the dermatophytes must scavenge for nutrients for growth, a process dependent on the induction of structural proteins, permeases and enzymes of the cell wall, in addition to the secretion of a variety of proteins and hydrolytic enzymes such as nucleases, lipases, non-specific proteases and keratinases that occur in response to a shortage in the supply of essential nutrients in the host. Dermatophytes de-repress non-specific proteolytic enzymes and keratinases which have optimum activity at acidic pH and are important virulence factors. Thus, their growth is dependent on the pH of the skin which being acidic gives an ideal ambient environment for the fungus. High transepidermal water loss values and impaired barrier function of the skin are correlated with high skin pH. Retinoid therapy is known to raise the skin pH, thereby possibly inhibiting dermatophyte growth.

Retinoids are generally thought to stimulate humoral and cellular immunity. They can enhance antibody production and stimulate peripheral blood T helper cells. Cell surface antigens of T cells and natural killer cells have been reported to increase after retinoid exposure in vitro. On the other hand, dermatophytes have mechanisms that allow them to evade the host response such as the immunosuppressive action of fungal mannans that causes reduction of inflammation and phagocytosis. Retinoids may counteract some of these immunosuppressive effects of the dermatophyte.

Finally, although more often associated with bacteria, pure fungal biofilms are a recognized entity, especially in yeasts like candida. Unlike candidal infections where the concept of fungal biofims has received considerable attention and is established, the same is not true for dermatophyte infections. Though it was introduced by Burkhart et al. to explain dermatophytomas, a form of onychomycosis refractory to standard antifungal therapies, it is a relatively virgin territory with hardly any published literature. The anecdotal efficacy of minocycline and isotretinoin in noninflammatory comedonal acne is more easily explained by their effects on altering the P acnes biofilm and lowering production of biological glue present in the biofilm. If the investigators can extrapolate the role of isotretinoin in P acnes biofilm to that of dermatophytes, it could potentially lead to tremendous insights into using an old but extremely efficacious drug for a novel indication.

Study design:

This will be a randomized open label single centre study. It will involve recruitment of patients with recurrent cutaneous dermatophytosis based on inclusion and exclusion criteria. The participants will be randomized (by block randomization) into four arms - Arm A will be treated with tablet terbinafine 250 mg once a day for 4 weeks, arm B will receive tablet terbinafine 250 mg once a day with low dose isotretinoin 20 mg/day, arm C will receive capsule itraconazole 200 mg/ day for 4 weeks, and arm D will be treated with capsule itraconazole 200 mg/ day for 4 weeks along with low dose isotretinoin (20 mg/day). Allocation concealment will be done by the sequentially numbered, opaque, sealed envelopes (SNOSE) method. After 4 weeks of treatment, arms B and D will continue to receive isotretinoin during subsequent 5 months of follow up.

Methodology All adults attending General OPD, Department of Dermatology, Venereology and Leprology, PGIMER, Chandigarh and satisfying the inclusion and exclusion criteria shall be eligible for recruitment in the present study after patients sign the written informed consent form. Complete physical examination including cutaneous, general and systemic examination will be done and recorded in case record proforma (annexure 1). Baseline clinical photographs will be taken for all patients.

ELIGIBILITY:
Inclusion Criteria:

• All patients with chronic recurrent dermatophytosis of more than 6 months duration who have been adequately treated for every episode still developing recurrences within one month of stopping oral antifungal drugs.

Exclusion Criteria:

* Patients with contraindications to receiving oral terbinafine, itraconazole or isotretinoin like those suffering from congestive cardiac failure, cardiac arrhythmias, liver or kidney function impairment or are on drugs whose plasma concentrations are likely to be increased by the concurrent administration of oral itraconazole.
* Pregnancy and lactation.
* Patients on immunosuppressive drugs.
* Immunocompromised patients (HIV positive/renal transplant etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
frequency of recurrences | 6 months
  The total number of patients who recur in the 4 different groups (comparing the paticipants who are on low dose isotretinoin during the follow up versus those who are not)

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Narang, MD, Principal Investigator — PGIMER CHANDIGARH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ardeshna KP, Rohatgi S, Jerajani HR. Successful treatment of recurrent dermatophytosis with isotretinoin and itraconazole. Indian J Dermatol Venereol Leprol. 2016 Sep-Oct;82(5):579-82. doi: 10.4103/0378-6323.183632. No abstract available. PMID 27297276